CLINICAL TRIAL: NCT07204236
Title: Study to Evaluate Immunogenicity and Safety of TVAX-008 Injection in Non/Treated Chronic Hepatitis B Patients With HBsAg≤20IU/ml or HBsAg Negative Without Serological Conversion
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Grand Theravac Life Sciences (Nanjing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YDSWX(TVAX-008)-004(IIT)
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TVAX-008 (Experimental): TVAX-008
  Interventions: Drug: TVAX-008

INTERVENTIONS:
Drug: TVAX-008 — TVAX-008

SUMMARY:
The objective of this study is to assess the immunogenicity and safety of TVAX-008 injection in antiviral untreated/untreated chronic hepatitis B patients with HBsAg≤20 IU/mL, or HBsAg negative and no seroconversion through an investigator-initiated clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18-65 years (inclusive);
2. Chronic hepatitis B patients with HBsAg<20 IU/mL without/on antiviral therapy; or HBsAg negative and no seroconversion population (HBsAg <20 IU/mL;HBVDNA<20 IU/mL; ）
3. HBsAg <10mIU/mL detected at least 4 weeks

Exclusion Criteria:

1. Use of immunosuppressants within 6 months prior to first dose:
2. Use of c1orticosteroids (other than topical or inhaled corticosteroids) for 1 week or more within 6 months prior to the first dose;
3. Hepatitis C virus (HCV), hepatitis D virus (HDV), Treponema pallidum (TP) antibody or human immunodeficiency virus (HIV) antibody positive:

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HBSAb levels after end of treatment | week24
  Change from baseline in HBSAb levels after end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Province Public Health Clinical Center, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No